CLINICAL TRIAL: NCT02593136
Title: Assessing Feasibility and Program Effectiveness of Home Fortification of Complementary Foods in Bihar: A Cluster Randomized Community Pilot
Brief Title: Home Fortification of Complementary Foods in Bihar India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Reynaldo Martorell, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00065311
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Anemia; Malnutrition
Keywords: Vitamins; Public Health; Nutrition
MeSH Terms: conditions — Anemia; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Fortification and Counseling (Experimental): Participants aged 6 to 18 months will receive a daily supplement of vitamins and minerals in dry powder form to be taken once daily for up to nine months or up to 240 sachets. Participant caregivers will also receive improved young child feeding practices (IYCF) counseling from a front line worker.
  Interventions: Dietary Supplement: Home Fortification Product (HFP); Other: Infant and Young Child Feeding (IYCF) Practices Counseling
- Improved Child Feeding Practices (IYCF) Counseling (Experimental): Participants ages 6 to 18 months will receive improved young child feeding practices (IYCF) counseling from a front line worker.
  Interventions: Other: Infant and Young Child Feeding (IYCF) Practices Counseling

INTERVENTIONS:
Dietary Supplement: Home Fortification Product (HFP) — The home fortification product (HFP) is a sachet containing multiple vitamins and nutrients as follows:
  Iron (Ferrous Fumarate) 12.5 mg Zinc (Zinc Gluconate) 5 mg Folic Acid 0.160 mg Vitamin-A (Vit-A Acetate) 0.30 mg Vitamin-C (Ascorbic Acid) 30 mg Vitamin-B12 0.9 mcg Iodine 90 mcg Maltodextrin (Base)
  Arms: Home Fortification and Counseling
Other: Infant and Young Child Feeding (IYCF) Practices Counseling — Infant and Young Child Feeding (IYCF) Practices Counseling provides direction on breast milk and milk feeding, food variety, and frequency for caregivers of children aged 6 to 18 months. Participants will be visited at least monthly by a field line worker for IYCF counseling and educational materials distribution.

SUMMARY:
This study evaluates the program effectiveness of home fortification along with infant and young child feeding (IYCF) counseling as a strategy to address anemia and complementary feedings gaps in a program setting of the Integrated Family Health Initiative being implemented by CARE India (a non-profit organization) in partnership with the Government of Bihar. The study also seeks to assess the field level worker experience with counseling and dissemination of home fortification products.

DETAILED DESCRIPTION:
This study evaluates the program effectiveness of home fortification along with infant and young child feeding (IYCF) counseling as a strategy to address anemia and complementary feedings gaps in a program setting of the Integrated Family Health Initiative being implemented by CARE India (a non-profit organization) in partnership with the Government of Bihar.The key objectives of this study are to examine acceptability and utilization by target population, assess impact on infant and young child feeding (IYCF) practices, evaluate impact on child growth, evaluate impact on hemoglobin concentration, and assess front line worker experience and motivation to disseminate enhanced counseling and home fortification products.

ELIGIBILITY:
Inclusion Criteria:

* Randomly selected children living within Health-Sub Centers (HSC) in West Champaran Bihar

Exclusion Criteria:

* Children less than six months of age
* Children greater than eighteen months of age

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11861 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of home fortification sachets consumed | Within 7 days (Up to 7 days)
  The number of sachets consumed versus those received by participants within seven days of distribution.
Number of home fortification sachets consumed | Within 31 days (Up to 31 days)
  The number of sachets consumed versus those received by participants within thirty one days of distribution.
Change in hemoglobin concentration | Baseline (month 0), Endline (month 12)
  Hemoglobin concentration will be collected by taking a small blood sample via finger or heal prick. A hemoglobin level below 7 g/dl is considered severe anemia.

SECONDARY OUTCOMES:
Frequency of home visits | Up to 12 months
  The number of times a front-line worker (FLW) visits one home within a twelve month period.
Frequency of home fortification sachet distribution | Up to twelve months
  The number of times a front-line worker (FLW) distributes home fortification sachets within a twelve month period.
Change in body length | Baseline (month 0), Endline (month 12)
  Child length will be measured using a SECA 417 length measuring board. Its measuring range is 10-100 cm with a graduation of 1 mm.
Change in body weight | Baseline (month 0), Endline (month 12)
  Child body weight will be measured using a SECA 874 mother-baby digital scale with capacity of 200 kg and graduation of 50 g < 150 kg > 100 g.
Complementary Feeding Rate | Month 6 (Up to six months)
  The percent of children initiating complementary feeding at six months.
Number of daily meals | Within 24 hours (Up to one day)
  The number of meals consumed per child in one day.
Quantity of food | Within 24 hours (Up to one day)
  The amount of food consumed by a child per meal in the home fortification and IYCF arm versus the IYCF alone arm.
Consistency of foods | Within 24 hours (Up to one day)
  The type of food textures (thick versus thin) consumed within 24 hours in the home fortification and IYCF arm versus the IYCF alone arm.
Diversity of foods | Within 24 hours (Up to one day)
  The number of different food groups consumed in one day in the home fortification and IYCF arm versus the IYCF alone arm.
Front-line worker motivation | Endline (Up to 9 months)
  Front-line worker (FLW) motivation to disseminate enhanced counseling and home fortification products will be measured at the end of study by the FLW survey. The FLW survey consists of questions regarding experience and perceived impact on work burden.
Change Developmental Milestones Checklist-II (DMC-II) | Baseline (month 0), Endline (month 12)
  Child development will be measured using the Developmental Milestones Checklist-II (DMC-II). The DMC-II is a 75-item parent report questionnaire evaluating gross motor, fine motor, language, personal-social skill development in children who are 3 to 24 months in age. The DMC-II has been slightly modified for this study by adding 7 items assessing cognitive development. The exact number of items administered depends on responses to previous items and the total range of score varies. Higher scores indicate increased development.
A-not-B task performance | Endline (month 12)
  Child executive function will be measured by direct child assessment using the A-not-B task in children 12-18 months of age only. Whether or not the child correctly identifies the location of a hidden toy is method of assessing development in early life.
Elicited imitation task performance | Endline (month 12)
  Child memory will be measured by direct child assessment using the Elicited imitation tasks in children 12-18 months of age only. Elicited imitation tasks are a tool to diagnose communication deficiencies in children. This test assesses whether or not a child can imitate the order of events of a sequence modeled by the evaluator.

CONTACTS AND LOCATIONS:
Overall Officials: Reynaldo Martorell, PhD, Principal Investigator — Emory University
Locations (1):
- CARE-India, Patna, Bihar, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keats EC, Das JK, Bhutta ZA. Micronutrient powders and diarrhoea risk in infants and young children - Authors' reply. Lancet Child Adolesc Health. 2021 Aug;5(8):e29-e30. doi: 10.1016/S2352-4642(21)00164-4. No abstract available. PMID 34302748
- [Derived] Larson LM, Young MF, Ramakrishnan U, Webb Girard A, Verma P, Chaudhuri I, Srikantiah S, Martorell R. A Cross-Sectional Survey in Rural Bihar, India, Indicates That Nutritional Status, Diet, and Stimulation Are Associated with Motor and Mental Development in Young Children. J Nutr. 2017 Aug;147(8):1578-1585. doi: 10.3945/jn.117.251231. Epub 2017 Jun 14. PMID 28615374